CLINICAL TRIAL: NCT06827756
Title: Comparative Study Between Norfloxacin, Nitazoxanide and Colistin As Secondary Prophylactic Agents for Spontaneous Bacterial Peritonitis
Brief Title: Comparative Study of Secondary Prophylaxis for SBP
Acronym: 3C-SPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dina Ahmed Esmat, Resident, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 33045/04/19
Record Dates: First submitted 2025-02-05; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Spontaneous Bacterial Peritonitis; Cirrhoses, Liver; Ascites
MeSH Terms: conditions — Ascites | interventions — Norfloxacin; nitazoxanide; Colistin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Norfloaxcin arm (Active Comparator): patients to receive norflxacin 400mg daily
  Interventions: Drug: Norfloxacin 400 MG
- Nitazoxaide arm (Active Comparator): patients to receive nitazoxaide 500mg daily
  Interventions: Drug: Nitazoxanide 500 MG
- Colisitn arm (Active Comparator): patients to receive Colistin 15 ml three times daily, totalling 2,25 MIU/ day
  Interventions: Drug: Colistin

INTERVENTIONS:
Drug: Norfloxacin 400 MG — Patients receiving Norfloxacin 400 Mg to prevent SBP
  Arms: Norfloaxcin arm
Drug: Nitazoxanide 500 MG — Patients receiving Nitazoxaide 500 Mg to prevent SBP
  Arms: Nitazoxaide arm
Drug: Colistin — Patients receiving Colistin 15ml three times/ day to prevent SBP
  Arms: Colisitn arm

SUMMARY:
The goal of this clinical trial is to learn if norfloxacin, nitazoxanide, and colistin work as secondary prophylactic agents for spontaneous bacterial peritonitis (SBP) in cirrhotic patients with ascites. It also aims to evaluate the safety and effectiveness of these treatments. The main questions it aims to answer are:

Are nitazoxanide and colistin as effective as norfloxacin in preventing recurrent SBP?

What medical outcomes do participants experience when taking norfloxacin, nitazoxanide, or colistin?

Researchers will compare norfloxacin, nitazoxanide, and colistin to determine their effectiveness in preventing SBP recurrence in cirrhotic patients.

Participants will:

Be randomly assigned to receive either 400 mg norfloxacin daily, 500 mg nitazoxanide twice daily, or 15 ml colistin syrup three times daily (2.25 MIU total per day).

Undergo regular blood tests and ascitic fluid analysis at discharge, 2 months, and 6 months post-treatment.

Be monitored for any side effects and recurrence of SBP.

ELIGIBILITY:
Inclusion Criteria:

Success Criteria: A ≥50% reduction in CRP within 3 months is considered a positive response.

* Ascitic patients diagnosed with Spontaneous Bacterial Peritonitis (SBP) by paracentesis.
* Ascitic fluid polymorphonuclear (PMN) cell count > 250/mm³.
* Age 50 years to 80 years.
* Willing to provide informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding females.
* History of allergic reactions to Norfloxacin, Nitazoxanide, or Colistin.
* Patients with recurrent spontaneous peritonitis.
* Presence of gastrointestinal hemorrhage.
* Renal failure (Creatinine > 2 mg/dL or on dialysis).
* Presence of severe infection-related sequelae (e.g., persistent fever, abdominal discomfort, sepsis).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Recurrence of Spontaneous Bacterial Peritonitis (SBP) | Baseline, 3 months, and 6 months
  Definition: The percentage of patients experiencing a recurrence of SBP within 6 months of treatment initiation.
  Measurement: Diagnosis confirmed by ascitic fluid analysis (PMN count > 250 cells/mm³ and positive culture).

SECONDARY OUTCOMES:
C-Reactive Protein (CRP) Reduction | Baseline, 1 month, 3 months, and 6 months
  Definition: A decrease in CRP levels, indicating a reduction in systemic inflammation.
  Measurement: CRP levels measured in mg/L.
  Success Criteria: A ≥50% reduction in CRP within 3 months is considered a positive response.
White Blood Cell (WBC) Count Reduction | Baseline, 1 month, 3 months, and 6 months
  Definition: Reduction in WBC count as a marker of infection control.
  Measurement: WBC count measured in x10³/µL.
  Success Criteria: A return to normal WBC count (<10,000/µL) by 3 months.
Renal Function Stability | Baseline, 3 months, and 6 months
  Definition: Prevention of renal impairment during treatment.
  Measurement: Serum Creatinine (mg/dL) and Blood Urea Nitrogen (BUN) (mg/dL).

OTHER OUTCOMES:
Adverse Events (Safety Assessment) | Throughout study duration (0-6 months)
  Definition: Frequency and severity of treatment-related side effects (e.g., diarrhea, nephrotoxicity, hypersensitivity reactions).
  Measurement: Patient-reported symptoms and clinical examination findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Faculty of Medicine, Tanta, Egypt